CLINICAL TRIAL: NCT01833611
Title: Phase IV Study of the Efficacy of Entecavir in Patients With Chronic Hepatitis B Virus Infection and Persistently Normal Alanine Aminotransferase
Brief Title: Entecavir for Chronic Hepatitis B Patients With Persistently Normal ALT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ting-Tsung Chang, Clinical Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ETV HR-96-23
Record Dates: First submitted 2012-04-27; First posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Hepatitis
MeSH Terms: conditions — Hepatitis, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETV group (Experimental): Entecavir 0.5mg at first year; then open with entecavir 0.5mg qd for 2nd, 3rd year
  Interventions: Drug: Entecavir
- Placebo group (Placebo Comparator): Placebo at first year, then opne with entecavir 0.5mg qd for 2nd, 3rd year
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Entecavir — entecavir 0.5mg qd
  Other Names: baraclude (generic name)
  Arms: ETV group
Drug: placebo — placebo qd
  Arms: Placebo group

SUMMARY:
Entecavir (ETV) has shown superior ability to suppress hepatitis B virus (HBV) replication, histology improvement as well as low rate of emergence of resistant mutants. Out of range of clinical recommendations for treatment of chronic hepatitis B (CHB), chronic HBV carriers with persistently normal ALT and viral load more than 10^5 copies/mL have progression of liver disease during long-term follow-up. In addition, certain proportions of these patients do have significant inflammation and fibrosis in liver histology. This study will be able to identify who are at risk of liver disease progression and evaluate efficacy of ETV regarding improvement of liver histology during short-term (1-year) and long-term ETV treatment (3-year).

DETAILED DESCRIPTION:
TITLE : A Randomized, Double-blind, Placebo-control Study Evaluating the Efficacy of Entecavir in Patients with Chronic Hepatitis B Virus Infection and Persistently Normal Alanine Aminotransferase INDICATION : Chronic hepatitis B virus infection with persistently normal ALT

OBJECTIVES :

Primary objective To evaluate the efficacy of entecavir (ETV) in improving liver histology in patients with chronic hepatitis B virus infection and persistently normal ALT.

The primary endpoint is to compare the proportion of subjects in each treatment group who achieve the histologic Endpoint, defined as improvement in the necroinflammatory score (≥ 2 point decrease in Knodell HAI score) and no worsening of fibrosis (≥ 1 point increase in the Knodell fibrosis score), at the Week 52 compared to baseline.

Secondary objectives

To compare the proportion of subjects in each treatment group with the following objectives at week 52, week 104, and week 156, and post-dosing 24 weeks:

1. Undetectable HBV DNA by the Roche TaqMan® HBV Test (limit of detection 60 IU/mL); HBV DNA by PCR will also be evaluated as a continuous parameter;
2. The reduction of HBV DNA from baseline.

STUDY DESIGN This is a 3-year prospective randomized, double-blind, placebo-control study. Enrolled subjects will be allocated according to HBeAg status (HBeAg-positive and HBeAg-negative), then randomized to ETV or placebo group.

ETV group: 1st year: ETV 0.5mg qd, then open with ETV 0.5mg qd for 2nd, 3rd year Placebo gr: 1st year: placebo, then open with ETV 0.5mg for 2nd, 3rd year

Dose of ETV: 0.5 mg/day Screening period: 6 weeks Timing of liver biopsy: baseline, 52th week, 156th week NUMBER OF PATIENTS 130 (1:1)

STUDY PERIOD NOV 2007 ~ MAY 2011 DRUG ADMINISTRAITON Route: oral Dose: ETV 0.5 mg/day Comparable placebo

STATISTICAL ANALYSIS Sample size determination:

An evaluation of the efficacy of entecavir compared to placebo is planned. A test for superiority of entecavir to placebo will be conducted that has high power to demonstrate superiority if there are larger histologic improvements of clinical importance. Histologic improvement after one year is estimated as 50% of entecavir treatment and 25% of placebo. Thus, a sample size of 47 will be required for 90% of confidence level with 5% of error. Finally, we estimate that it will be appropriate to enroll 65 patients in each arm due to probably patients' withdrawal.

Statistical Analyses The difference in response rates for the Histologic Endpoint (entecavir-placebo) along with its standard error and 95% confidence interval will be computed. Subset analyses defined by prognostic variables [e.g. gender, and HBV DNA level] for the Histologic Endpoint will be performed.

Change from baseline at Week 52 and 156 in Knodell Scores will also be summarized as a continuous parameter. The secondary efficacy variables will also be summarized and compared between the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged between 18 and 65 year-old with history of chronic hepatitis B virus infection;
2. Detectable HBsAg at screening and for at least 24 weeks prior to screening or detectable HBsAg for < 24 week and negative for IgM core antibody and confirmation of chronic hepatitis on liver biopsy;
3. ALT should be within normal range in recent one year and at least twice, which are at least 3 month apart;
4. Normal ALT at screening;
5. Screening HBV DNA of more than 10^5 copies/mL by Roche AmplicorTM PCR assay performed by the central laboratory;
6. Evidence of chronic hepatitis on liver biopsy (Knodell HAI Score >= 4) performed ≤ 52 weeks prior to randomization;
7. All women of childbearing potential must have a negative serum or urine pregnancy test.

Exclusion Criteria:

1. Coinfection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis D virus (HDV);
2. Other forms of liver disease e.g., alcoholic, autoimmune, biliary disease;
3. Patients with evidence of decompensation of liver disease;
4. Therapy with interferon, thymosin alpha or antiviral agents with activity against hepatitis B (e.g., adefovir, famciclovir, lamivudine, and telbivudine) within 24 weeks of randomization into this study;
5. More than 12 weeks of prior therapy with nucleoside or nucleotide analogue antiviral agents with activity against hepatitis B (e.g., adefovir, famciclovir lamivudine, and telbivudine);
6. Prior therapy with entecavir;
7. Known history of allergy to nucleoside analogues;
8. Hemoglobin < 10.0 g/dL;
9. Platelet count < 75,000/mm3;
10. Absolute neutrophil count< 1500 cells/mm3;
11. Creatinine > 1.5mg/dL (133 μmol/L);
12. Anti-nuclear antibody (ANA) titer > l :160 unless attributable to non-hepatic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2008-09; Primary Completion 2014-11 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of liver histology in patients with chronic hepatitis B virus infection and persistently normal ALT receiving entecavir. Please refer to "Description" section for the definiton of improvement of liver histology | 1 year
  1. The ratio of liver histology improvement in two groups.
  2. Definition of improving liver histology is improvement in the necroinflammatory score (≥ 2 point decrease in Knodell necroinflammation score) and no worsening of fibrosis (≥ 1 point increase in the Knodell fibrosis score) at the week 52 liver biopsy compared to baseline.

SECONDARY OUTCOMES:
Undetectable HBV DNA | 1 year and 3 year
  1. The ratio of undetectable HBV DNA in two groups
  2. HBV DNA by the Roche TaqMan® HBV Test (limit of detection 60 IU/mL)
the reduction of HBV DNA from baseline | 1 year and 3 year
  1. expressed with Log 10 coipes/ml
  2. HBV DNA by the Roche TaqMan® HBV Test (limit of detection 60 IU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Tsung Chang, MD. PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (4):
- Taiwan (4):
  - Buddhist Dalin Tzu-Chi General Hospital, Chiayi City
  - Chia-Yi Christian Hospital, Chiayi City
  - Chang-Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City

REFERENCES:
- [Derived] Tseng KC, Chen CY, Tsai HW, Chang TT, Chuang WL, Hsu PI, Liu WC, Cheng PN. Efficacy of entecavir in chronic hepatitis B patients with persistently normal alanine aminotransferase: randomized, double-blind, placebo-controlled study. Antivir Ther. 2014;19(8):755-64. doi: 10.3851/IMP2754. Epub 2014 Feb 28. PMID 24583931